CLINICAL TRIAL: NCT03813524
Title: Early Feasibility Study of the Cardiovalve Transfemoral Mitral Valve System
Brief Title: Cardiovalve Transfemoral Mitral Valve System
Acronym: AHEAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID Impact
Sponsor: Boston Biomedical Associates (Other)
Collaborators: Cardiovalve Ltd. (Industry); Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 18-01
Record Dates: First submitted 2019-01-16; First posted 2019-01-23 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Cardiovalve Transfemoral Mitral Valve (Experimental): Replacement valve delivered through a transfemoral access and transseptal approach
  Interventions: Device: Cardiovalve Transfemoral Mitral Valve

INTERVENTIONS:
Device: Cardiovalve Transfemoral Mitral Valve — The Cardiovalve Transfemoral Mitral Valve System is intended for use symptomatic patients with severe mitral regurgitation who are at elevated risk for surgical mitral valve repair or replacement and who are anatomically eligible for transfemoral mitral valve replacement with transseptal access to the left atrium.

SUMMARY:
This study is to evaluate the safety and technical performance of the Cardiovalve Transfemoral Mitral Valve System with its associated procedure, to minimize mitral regurgitation. Data collected in this clinical study will include 30-day safety and performance of the device and delivery system, and long-term clinical outcomes over a follow-up of 5 years.

DETAILED DESCRIPTION:
The Cardiovalve offers a replacement valve delivered through a transfemoral access and transseptal approach, and is intended to reduce mortality and adverse event rates in selected patients for whom surgical options are not feasible.

Innovation: A truly transfemoral, trans venous delivery of the valve which minimizes procedural risk. The Cardiovalve implant has a very low left ventricle (LV) protrusion footprint thus reducing the risk of LV outflow tract obstruction and/or interference with the LV. The experience to date is limited but thus far none of the clinical programs has been halted for safety reasons. Most of the technologies have focused on a transapical delivery approach (with mini-thoracotomy access) to further simplify the delivery method, with only a few allowing trans-septal delivery with femoral venous access.

ELIGIBILITY:
Inclusion Criteria:

* 85>Age ≥ 18 years
* Symptomatic (Stage D) severe MR confirmed by the echo core lab
* Cardiac Index > 2.0
* Left Ventricular Ejection Fraction (LVEF) is ≥ 30% (within 90 days prior to subject enrollment based upon TTE)
* New York Heart Association (NYHA) Functional Class II, III or ambulatory IVa
* Prior treatment with Guideline Directed Medical Therapy (GDMT) for heart failure for at least 30 days prior to index procedure
* Patient deemed a high surgical risk per MVARC definition by the site's Heart Team (as a minimum, one MV cardiac surgeon and one interventional cardiologist, and a cardiac imaging expert).

Exclusion Criteria:

* MR etiology that is exclusively Primary (degenerative)
* Echocardiographic or angiographic evidence of severe mitral annular calcification
* Echocardiographic evidence of EROA < 0.3cm2
* Untreated clinically significant coronary artery disease requiring revascularization.
* Hypertrophic/restrictive cardiomyopathy, constrictive pericarditis, or other structural heart disease causing heart failure other than other than cardiomyopathy of either ischemic or non-ischemic etiology
* Hypotension (systolic pressure < 90 mm Hg)/Cardiogenic shock or other hemodynamic instability requiring the need for inotropic
* Fixed pulmonary artery systolic pressure > 2/3 of systemic systolic blood pressure
* LVEDD >75 mm
* Severe tricuspid regurgitation or evidence of severe right ventricular dysfunction.
* Anatomy deemed not suitable for the Cardiovalve
* Elevated Creatine Kinase-MB (CK-MB)
* UNOS Status 1 heart transplant or prior orthotropic heart transplantation.
* Life Expectancy < 1 year due to non-cardiac conditions
* NYHA functional class IVb
* Chronic Kidney Disease with Creatinine clearance <30 ml/min/1.73m2
* Any prior mitral valve surgery or transcatheter mitral valve procedure
* Stroke or transient ischemic event within 30 Days prior to index procedure
* Modified Rankin Scale > 4 disability
* Class I indication for biventricular pacing (in patient with CRT device not implanted)
* Implant or revision of any rhythm management device (CRT or CRT-D) or implantable cardioverter-defibrillator within one month prior to index procedure
* Need for cardiovascular surgery (other than MV disease)
* Echocardiographic evidence of intracardiac mass, thrombus, or vegetation
* Active endocarditis
* Known severe symptomatic carotid stenosis (> 70 % via ultrasound)
* Active infections requiring current antibiotic therapy
* Active cancer with expected survival < one year
* Pregnant or planning pregnancy within next 12 months.
* Currently participating in an investigational drug or another device study
* Any condition making it unlikely the patient will be able to complete all procedures
* Patient (or legal guardian) unable or unwilling to provide written, informed consent before study enrollment
* Subjects in whom transesophageal echocardiography is contraindicated
* Known hypersensitivity or contraindication to procedural, post procedural medication (e.g., contrast solution, heparin, anticoagulation therapy) or hypersensitivity to nickel or titanium.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Cardiovalve Technical Success | 30 Days
  1. Successful access, delivery and retrieval of the delivery system; and
  2. Successful deployment and correct positioning of the first intended implant; and
  3. Freedom from emergency surgery or reintervention related to the device or access procedure
  Without any procedural mortality, stroke, and device dysfunction (Central MR grade > 1 or paravalvular leak moderate or severe, mean mitral gradient > 6 mm Hg, LVOT obstruction (gradient increase ≥10 mm Hg)) at 30-day follow up.
Cardiovalve to be implanted without Major Device Related Adverse Events through 30 Days including: | 30 Days
  1. Death (Cardiovascular mortality vs non-cardiovascular);
  2. Reintervention (operative or transcatheter) due to progressive or recurrent MR or device related complications;
  3. Disabling Stroke;
  4. Myocardial infarction (MVARC definition);
  5. Major access site and vascular complications
  6. Fatal or Life-threatening bleeding (MVARC Type III- V)
  7. Life-threatening arrhythmia;
  8. Renal Failure requiring dialysis;

SECONDARY OUTCOMES:
Mitral Regurgitation severity | 30 days, 3 months, 6 months
Change in LV end diastolic volume index (LVEDVI) | 30 days, 3 months, 6 months
Change in LV end systolic volume index (LVESVI) | 30 days, 3 months, 6 months
Changes in New York Heart Association (NYHA) functional class | 30 days, 3 months, 6 months
  Class I-IV; Higher functional class represents more severe symptoms of heart failure
6-minute walk test (6MWT) distance | 30 days, 3 months, 6 months
Kansas City Cardiomyopathy Questionnaire (KCCQ) score | 30 days, 3 months, 6 months
  3 subscales: Symptom Burden- range 0-100; Physical Limitation- range 0-100; Quality of Life- range 0-100;
  Higher score represents less burdensome symptoms within each subscale. The total KCCQ score represents the mean (average) of the three subscale scores.
Clinical Frailty Score | 30 days, 3 months, 6 months
  Scale from 1 to 9 Lower score indicates a lower level of frailty

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Piedmont Heart Institute, Atlanta, Georgia
  - Columbia University Medical Center/NYPH, New York, New York

IPD SHARING:
Plan to Share IPD: No